CLINICAL TRIAL: NCT00104416
Title: A Multicenter, Double-blind, Randomized, Parallel-group Evaluation of LAMICTAL Extended-Release Adjunctive Therapy in Patients With Primary Generalized Tonic-Clonic Seizures
Brief Title: Study Evaluating LAMICTAL Extended-Release Therapy Added To Current Seizure Treatments In Patients With Primary Generalized Tonic-Clonic Seizures (PGTC) Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LAM100036
Record Dates: First submitted 2005-02-28; First posted 2005-03-01 (Estimated); Results first posted 2010-05-18 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-11

CONDITIONS: Epilepsy, Tonic-Clonic
Keywords: antiepileptic drugs; seizures; primary generalized tonic-clonic seizures; Epilepsy; lamotrigine; anticonvulsants; LAMICTAL
MeSH Terms: conditions — Epilepsy, Tonic-Clonic; Seizures; Epilepsy | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- lamotrigine (LAMICTAL) extended-relesase (Experimental)
  Interventions: Drug: lamotrigine (LAMICTAL) extended-release

INTERVENTIONS:
Drug: lamotrigine (LAMICTAL) extended-release — Primary experimental dosage form
  Arms: lamotrigine (LAMICTAL) extended-relesase
Drug: Placebo — Placebo control
  Arms: Placebo

SUMMARY:
This study is being conducted to compare the efficacy and safety of LAMICTAL (lamotrigine) extended-release with placebo in the treatment of Primary Generalized Tonic-Clonic (PGTC) seizures. LAMICTAL extended-release is an investigational drug. Placebo tablets look like LAMICTAL extended-release tablets but do not contain active medication. In this study, LAMICTAL extended-release or placebo tablets will be added to current seizure treatments.

ELIGIBILITY:
Inclusion Criteria:

* Is ≥13 years of age (male or female).
* Has a confident diagnosis of epilepsy with PGTC seizures for more than 24 weeks prior to the Baseline Phase.
* Has electroencephalogram (EEG) evidence of either spike-and-wave discharges consistent with PGTC, or at least 2 EEGs with no indication of focal abnormalities. The EEG may be historical or prospective. Investigators may use a historical EEG as long as there is appropriate documentation.
* Has a documented history of PGTC seizures with or without other generalized seizure type(s) with no focal onset, and at least 1 PGTC seizure during the eight consecutive weeks (i.e., 56 consecutive days) prior to starting the 8-week Baseline Phase.
* Has at least 3 PGTC seizures occurring anytime during an 8-week (i.e., 56 days) prospective Baseline Phase.

  * NOTE: When a historical baseline is used, the same time period cannot count for documentation of inclusion criteria 4 and 5. Additionally, innumerable seizure activity will not count towards the number of seizures required for randomization.
  * NOTE: With authorization from GSK, a maximum of four weeks (i.e., 28 days) of historical seizure data may replace up to four weeks (i.e., 28 days) of the prospective Baseline Phase for subjects providing reliable documentation of the following:

    1. complete daily seizure diary that includes the number of seizures experienced each day along with the exact classification of each seizure type for consecutive days prior to the prospective Baseline Phase
    2. stability of prescribed dosages of background antiepileptic drugs (AEDs)
    3. compliance with background AEDs.
  * All subjects permitted to use historical seizure data must complete a minimum of four weeks (i.e., 28 days) of the prospective Baseline Phase. The historical Baseline Phase and the prospective Baseline Phase must equal 56 consecutive days.
* Is currently treated with a stable regimen of one or two AED(s) for at least four weeks prior to starting the Baseline Phase (historical or prospective).

  * NOTE: Benzodiazepines used chronically will be considered to be concurrent AEDs.
  * NOTE: Subjects with surgically implanted vagal nerve stimulators (VNS) will be allowed to enter the study provided that all of the following conditions are met:

    1. VNS has been in place for at least 24 weeks prior to the Baseline Phase.
    2. The settings must remain the same for at least 28 days prior to the Baseline Phase.
    3. The settings must remain the same during the Baseline, Escalation, Maintenance and Transition Phases.
    4. The battery is expected to last for the duration of the study.
    5. VNS is counted as a "concurrent AED."
* Is able and willing to maintain an accurate and complete daily written seizure diary, or has a parent/caregiver who is able and willing to maintain an accurate and complete daily written seizure diary for the entire duration of the study.
* Is able to comply with dosing of study drugs, background AEDs and all study procedures.
* Has given written informed consent, or has a parent/legally authorized representative who has given written informed consent, prior to the performance of any study assessments.
* If female, and of childbearing potential, must be using an acceptable form of birth control, to include one of the following:

  1. Complete abstinence from intercourse for two weeks before exposure to the study drug, throughout the clinical trial, and for a period after the trial to account for elimination of the drug (a minimum of 3 weeks).
  2. Consistent and correct use of one of the following methods of birth control:

     * Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject
     * Implants of levonorgestrel
     * Injectable progestogen
     * Oral contraceptive (either combined, with at least 50mcg estrogen for women on enzyme-induced AEDs, or progestogen only)
     * Any intrauterine device (IUD) with a documented failure rate of less than 1% per year
     * Double barrier method consisting of spermicide plus a mechanical barrier (e.g., spermicide plus a male condom or a female diaphragm).
     * NOTE: Women who have had a hysterectomy, tubal ligation, or are post-menopausal are considered to be of non-childbearing potential.

Exclusion Criteria:

* Has a history of partial seizures or interictal expression of partial seizures as evidenced by EEG NOTE: EEG may be historical or prospective.
* Has had status epilepticus within the 24 weeks prior to, or during, the Baseline Phase.
* Is taking three or more background AEDs chronically.
* Has Lennox-Gastaut syndrome.
* Is currently using or has previously used lamotrigine.
* Is currently taking felbamate.
* Is abusing alcohol and/or other substance(s).
* Has taken an investigational drug within the previous 30 days or plans to take an investigational drug anytime during the study.
* Is receiving chronic treatment with any medication that could influence seizure control. NOTE: Use of benzodiazepines is allowed.
* Is currently following the ketogenic diet.
* Is planning surgery to control seizures during the study.
* Is suffering from acute or progressive neurological disease, severe psychiatric disease, or severe mental abnormality that are likely to interfere with the objectives of the study.
* Has any clinically significant cardiac, renal, hepatic condition, or a condition that affects the absorption, distribution, metabolism or excretion of drugs.
* Is pregnant, breastfeeding, or planning to become pregnant during the study or within the three weeks after the last dose of study drug.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2004-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (118):
- United States (59):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Northport, Alabama
  - GSK Investigational Site, Tuscaloosa, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Sepuldeva, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Maitland, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Suwanee, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Flossmoor, Illinois
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Crestview Hills, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Traverse City, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Edison, New Jersey
  - GSK Investigational Site, West Orange, New Jersey
  - GSK Investigational Site, Amherst, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Wichita Falls, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Burlington, Vermont
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
- Argentina (2):
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, Buenos Aires
- Brazil (3):
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, Campinas, São Paulo
  - GSK Investigational Site, São Paulo, São Paulo
- GSK Investigational Site, Santiago, Región Metro de Santiago, Chile
- Germany (37):
  - GSK Investigational Site, Singen, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Alzenau in Unterfranken, Bavaria
  - GSK Investigational Site, Bamberg, Bavaria
  - GSK Investigational Site, Fürth, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Neuötting, Bavaria
  - GSK Investigational Site, Straubing, Bavaria
  - GSK Investigational Site, Unterhaching, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Bernau bei Berlin, Brandenburg
  - GSK Investigational Site, Ludwigsfelde, Brandenburg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Bad Homburg, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Bückeburg, Lower Saxony
  - GSK Investigational Site, Göttingen, Lower Saxony
  - GSK Investigational Site, Osnabrück, Lower Saxony
  - GSK Investigational Site, Wismar, Mecklenburg-Vorpommern
  - GSK Investigational Site, Baesweiler, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Hattingen, North Rhine-Westphalia
  - GSK Investigational Site, Mönchengladbach, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Limburgerhof, Rhineland-Palatinate
  - GSK Investigational Site, Flöha, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Bernburg, Saxony-Anhalt
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Köthen, Saxony-Anhalt
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Naumburg, Saxony-Anhalt
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Jena, Thuringia
- India (3):
  - GSK Investigational Site, Hyderabad, Andhra Pradesh
  - GSK Investigational Site, Lucknow
  - GSK Investigational Site, New Delhi
- GSK Investigational Site, Kubang Kerian, Malaysia
- Puerto Rico (2):
  - GSK Investigational Site, San Germán, Puerto Rico
  - GSK Investigational Site, San Juan, Puerto Rico
- Russia (5):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, St'Petersburg
  - GSK Investigational Site, Yekaterinburg
- South Korea (2):
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Seoul
- Ukraine (3):
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lviv

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Biton V, Di Memmo J, Shukla R, Lee YY, Poverennova I, Demchenko V, Saiers J, Adams B, Hammer A, Vuong A, Messenheimer J. Adjunctive lamotrigine XR for primary generalized tonic-clonic seizures in a randomized, placebo-controlled study. Epilepsy Behav. 2010 Nov;19(3):352-8. doi: 10.1016/j.yebeh.2010.07.022. Epub 2010 Oct 30. PMID 20937567
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: LAM100036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LAM100036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: LAM100036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: LAM100036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: LAM100036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: LAM100036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: LAM100036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants (par.) that complete the Treatment Phase (TP) and all Baseline Failures (par. who did not meet randomization seizure criteria necessary to qualify for the TP) are eligible to enter the Continuation Phase (CP). The CP is for long-term safety exposure to lamotrigine (LTG) extended release (XR); it is not a cross-over phase.
Pre-assignment Details: The number of par. starting the CP does not equal the number completing the TP, as 1) the CP was optional, 2) not everyone from the TP was eligible to enter the CP, and 3) Baseline Failures were allowed to enter the CP, however they were not included in the "started" count for the TP.
Groups:
- Double-Blind Phase: Placebo: Control - matching placebo once daily
- Double-Blind Phase: LTG XR: Lamotrigine (LTG) extended release (XR) once daily
- Continuation Phase: Placebo/LTG: Participants who received placebo in the Double-Blind Phase and then entered the CP, in which they received LTG
- Continuation Phase: LTG/LTG: Participants who received LTG XR in the Double-Blind Phase and then entered the CP, in which they received LTG
- Baseline Failures: Baseline failures who entered the CP without receiving treatment in the Double-Blind Phase. Baseline Failures were participants that successfully progressed through the Screening Phase and completed the Baseline Phase of the Double-blind Study, but ultimately did not meet the seizure frequency criteria for randomization into the Double-Blind Treatment Phase of the study. As a result, they were not counted as having started in the Double-Blind Study, but were eligible to enter the CP of the study.
Period: Double-Blind Phase
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: LTG XR | Continuation Phase: Placebo/LTG | Continuation Phase: LTG/LTG | Baseline Failures
Started | 77 | 76 | 0 | 0 | 0
Completed | 69 | 66 | 0 | 0 | 0
Not Completed | 8 | 10 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0
Not completed — Participant Did Not Take Drug | 3 | 4 | 0 | 0 | 0
Period: Continuation Phase
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: LTG XR | Continuation Phase: Placebo/LTG | Continuation Phase: LTG/LTG | Baseline Failures
Started | 0 | 0 | 69 | 67 (One participant did not complete the Double-Blind Phase but was enrolled in the Continuation Phase.) | 32
Completed | 0 | 0 | 63 | 65 | 27
Not Completed | 0 | 0 | 6 | 2 | 5
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1 | 1
Not completed — Pregnancy | 0 | 0 | 1 | 1 | 0
Not completed — Non-compliance | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Double-Blind Phase: LTG XR: LTG XR once daily
- Total: Total of all reporting groups
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: LTG XR | Total
Number analyzed (Participants) | 73 | 70 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline measures are on the Intent-to-Treat (ITT) Population, participants who took at least 1 dose of study drug and had at least 1 post-baseline efficacy assessment. Four and six participants did not meet the ITT definition in the Double-Blind Treatment Phase Placebo Arm and the Double-Blind Treatment Phase LTG XR Arm, respectively.
  years | 28.4 (11.48) | 29.4 (12.78) | 28.9 (12.10)
Gender [Count of Participants; unit: Participants] — Baseline measures are on the Intent-to-Treat (ITT) Population, participants who took at least 1 dose of study drug and had at least 1 post-baseline efficacy assessment. Four and six participants did not meet the ITT definition in the Double-Blind Treatment Phase Placebo Arm and the Double-Blind Treatment Phase LTG XR Arm, respectively.
  Participants
    Female | 38 | 32 | 70
    Male | 35 | 38 | 73
Race/Ethnicity, Customized [Number; unit: participants] — Baseline measures are on the Intent-to-Treat (ITT) Population, participants who took at least 1 dose of study drug and had at least 1 post-baseline efficacy assessment. Four and six participants did not meet the ITT definition in the Double-Blind Treatment Phase Placebo Arm and the Double-Blind Treatment Phase LTG XR Arm, respectively.
  participants
    African American/African Heritage | 1 | 2 | 3
    Asian | 31 | 31 | 62
    White | 38 | 37 | 75
    American Indian or Alaskan Native and White | 2 | 0 | 2
    Asian and White | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Weekly Primary Generalized Tonic-clonic (PGTC) Seizure Frequency During the Entire Double-Blind Treatment Phase
Description: Percent change from baseline is calculated as the number of seizures by week during the Double-Blind Treatment Phase (Treatment Week 1 up to Week 19) compared to the number of seizures per week during the Baseline Phase (Baseline Week 1 up to Week 8). A positive number equals a reduction in seizure frequency. PGTC seizures are more commonly known as gran mal seizures.
Time Frame: Baseline through end of Double-Blind Treatment Phase (up to Week 19)
Population: Intent-to-Treat (ITT) Population: all randomized participants who took at least one dose of study drug and had at least one post-baseline efficacy assessment in the Double-Blind Treatment Phase. One participant in each treatment group did not have any PGTC seizures during the Baseline Phase.
Measure: Median (Full Range); unit: percent change
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: LTG XR
Number analyzed (Participants) | 72 | 69
percent change | 32.1 [-427 to 100] | 75.4 [-100 to 100]
Statistical Analysis 1: Comparison: Double-Blind Phase: Placebo vs Double-Blind Phase: LTG XR; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Median Difference (Final Values) = 31.6, 95% CI [15.8 to 48.1]

2. Secondary Outcome: Number of Participants With >=25%, >=50%, >=75%, or 100% Reduction in PGTC Seizure Frequency During the Entire Double-Blind (DB)Treatment Phase (TP), the Escalation Phase, the Maintenance Phase, and the Last 8 Weeks of the Maintenance Phase
Description: Change in seizure frequency was calculated as the average seizure frequency during each of the following: the Entire DB Treatment Phase (Treatment Week 1 up to Week 19); the Escalation Phase (Treatment Week 1 up to Week 7); the Maintenance Phase (Treatment Week 8 up to Week 19); and the last 8 weeks of the Maintenance Phase (Treatment Week 12 up to Week 19), minus the seizure frequency at Baseline.
Time Frame: Entire DB Treatment Phase (Treatment Week 1 up to Week 19), Escalation Phase (Treatment Week 1 up to Week 7), Maintenance Phase (Treatment Week 8 up to Week 19), and the last 8 weeks of the Maintenance Phase (Treatment Week 12 up to Week 19)
Population: ITT Population. One participant in each treatment group did not have any PGTC seizures during the Baseline Phase, as a result they were not counted in this efficacy endpoint; an additional 2 and 1 participants in the Placebo and LTG XR group, respectively, were not counted in the Maintenance Phase (MP) or last 8 weeks of MP due to study withdrawal.
Measure: Number; unit: participants
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: LTG XR
Number analyzed (Participants) | 72 | 69
participants
  >=25% reduction, Entire DB TP, n=72, 69 | 43 | 56
  >=50% reduction, Entire DB TP, n=72, 69 | 23 | 48
  >=75% reduction, Entire DB TP, n=72, 69 | 14 | 35
  100% reduction, Entire DB TP, n=72, 69 | 7 | 14
  >=25% reduction, Escalation Phase, n=72, 69 | 39 | 51
  >=50% reduction, Escalation Phase, n=72, 69 | 23 | 38
  >=75% reduction, Escalation Phase, n=72, 69 | 14 | 24
  100% reduction, Escalation Phase, n=72, 69 | 9 | 15
  >=25% reduction, Maintenance Phase, n=70, 68 | 46 | 60
  >=50% reduction, Maintenance Phase, n=70, 68 | 29 | 51
  >=75% reduction, Maintenance Phase, n=70, 68 | 14 | 40
  100% reduction, Maintenance Phase, n=70, 68 | 10 | 31
  >=25% reduction, Last 8 Weeks of MP, n=70, 68 | 47 | 61
  >=50% reduction, Last 8 Weeks of MP, n=70, 68 | 29 | 54
  >=75% reduction, Last 8 Weeks of MP, n=70, 68 | 18 | 44
  100% reduction, Last 8 Weeks of MP, n=70, 68 | 15 | 35

3. Secondary Outcome: Percent Change From Baseline in PGTC Seizure Frequency During the Escalation Phase, the Maintenance Phase, and During the Last 8 Weeks of the Maintenance Phase of the Double-Blind Treatment Phase
Description: Percent change from baseline is calculated as the number of seizures by week during the Escalation Phase (Treatment Week 1 up to Week 7), the Maintenance Phase (Treatment Week 8 up to Week 19), and during the last 8 weeks of the Maintenance Phase (Treatment Week 12 up to Week 19) compared to the number of seizures per week during the Baseline Phase (Baseline Week 1 up to Week 8). A positive number equals a reduction in seizure frequency.
Time Frame: Escalation Phase (Treatment Week 1 up to Week 7), Maintenance Phase (Treatment Week 8 up to Week 19), and the last 8 weeks of the Maintenance Phase (Week 12 up to Week 19)
Population: ITT Population. One participant in each treatment group did not have any PGTC seizures during the Baseline Phase as a result they were not counted for this efficacy endpoint; an additional 2 and 1 participants in the Placebo and LTG XR group, respectively, were not counted in the Maintenance Phase (MP) or last 8 weeks of MP due to study withdrawal.
Measure: Median (Full Range); unit: percent change
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: LTG XR
Number analyzed (Participants) | 72 | 69
percent change
  Escalation Phase, n=72, 69 | 30.6 [-319 to 100] | 61.9 [-197 to 100]
  Maintenance Phase, n=70, 68 | 33.3 [-492 to 100] | 89.7 [-142 to 100]
  Last 8 weeks of the Maintenance Phase, n=70, 68 | 35.4 [-180 to 100] | 100.0 [-131 to 100]

4. Secondary Outcome: Number of Participants With the Indicated Time to >=50% Reduction in Seizure Frequency in the Double-Blind Treatment Phase
Description: 50% reduction in seizure frequency is defined as the time at which a participant first achieved and maintained a >=50% reduction in seizure frequency following exposure to at least 1 week of study drug.
Time Frame: Baseline through end of Double-Blind Treatment Phase (up to Week 19)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: LTG XR
Number analyzed (Participants) | 73 | 70
participants
  2 weeks | 12 | 22
  4 weeks | 12 | 28
  8 weeks | 14 | 39
  12 weeks | 20 | 43
  16 weeks | 23 | 48

5. Secondary Outcome: Change From Baseline in Body Weight at Week 19 of the Double-Blind Treatment Phase
Description: Change from baseline in body weight is calculated as the Week 19 (or last on-study measurement in Double-Blind Treatment Phase) value minus the Baseline value.
Time Frame: Baseline and Week 19 (or last on-study measurement in Double-Blind Treatment Phase)
Population: ITT Population
Measure: Median (Full Range); unit: kilograms
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: LTG XR
Number analyzed (Participants) | 73 | 70
kilograms | 1.00 [-7.7 to 10.0] | 0.00 [-11.4 to 8.8]

6. Secondary Outcome: Number of Participants With Improved Clinical Status on the Investigator's Global Assessment in the Double-Blind Treatment Phase
Description: The investigators rated the participants' overall clinical status based on 7 clinical factors and an overall factor: seizure frequency, duration, and intensity; adverse experiences; social, intellectual, and motor functioning. Using a 7-point scale (marked deterioration [1], moderate deterioration [2], mild deterioration [3], no change [4], mild improvement [5], moderate improvement [6], or marked improvement [7]), the investigators assessed the participants' status compared to their condition prior to initiating study medication.
Time Frame: Week 19 (or last on-study assessment in Double-Blind Treatment Phase)
Population: ITT Population. Overall clinical status not assessed for 2 participants in each of the Placebo and LTG XR groups, respectively.
Measure: Number; unit: participants
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: LTG XR
Number analyzed (Participants) | 71 | 68
participants
  Any improvement, score of 5-7 | 36 | 57
  No change, score of 4 | 33 | 10
  Any deterioration, score of 1-3 | 2 | 1

7. Secondary Outcome: Number of Participants With Improved Satisfaction With Seizure Control on the Subject Satisfaction Questionnaire in the Double-Blind Treatment Phase
Description: Participants were asked to rate their satisfaction with their seizure control compared to their seizure control prior to initiating study drug on a 7 point scale: marked deterioration (1), moderate deterioration (2), mild deterioration (3), no change (4), mild improvement (5), moderate improvement (6), or marked improvement (7).
Time Frame: Week 19 (or last on-study assessment in Double-Blind Treatment Phase)
Population: ITT Population. Participant satisfaction was not assessed for 2 participants in each of the Placebo and LTG XR groups, respectively.
Measure: Number; unit: participants
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: LTG XR
Number analyzed (Participants) | 71 | 68
participants
  Any improvement, score of 5-7 | 53 | 60
  No change, score of 4 | 13 | 6
  Any deterioration, score of 1-3 | 5 | 2

8. Secondary Outcome: Percent Change From Baseline in Weekly PGTC Seizure Frequency During the Entire Continuation Phase (CP), the Transition Phase, the Open-Label Phase, and the Last 8 Weeks of the Open-Label Phase
Description: Percent change from baseline is calculated as the number of seizures by week during the entire CP (CP Week 1 up to Week 52), the Transition Phase (CP Week 1 up to Week 7), the Open-Label Phase (CP Week 8 up to Week 52), and the last 8 weeks of the Open-Label Phase (CP Week 45 up to Week 52) minus the number of seizures per week during the Baseline Phase (Baseline Week 1 through Week 8). A positive number equals a reduction in seizure frequency.
Time Frame: Entire CP (CP Week 1 up to Week 52), the Transition Phase (CP Week 1 up to Week 7), the Open-Label Phase (CP Week 8 up to Week 52), and the last 8 weeks of the Open-Label Phase (CP Week 45 up to Week 52)
Population: ITT Population for CP: all participants who took at least one dose of study medication during the CP and had at least one post baseline seizure assessment during the CP. Variability in participant numbers are due to not having any PGTC seizures during the Baseline Phase and study withdrawal prior to progressing to the next phase.
Measure: Median (Full Range); unit: percent change
Groups:
- Continuation Phase: Placebo/LTG: Placebo participants who entered the CP
- Continuation Phase: LTG/LTG: LTG XR participants who entered the CP
- Baseline Failures: Baseline failures who entered the CP
Arm/Group | Continuation Phase: Placebo/LTG | Continuation Phase: LTG/LTG | Baseline Failures
Number analyzed (Participants) | 68 | 66 | 24
percent change
  Entire Continuation Phase, n=68, 66, 24 | 85.2 [-113.3 to 100.0] | 95.1 [-100.0 to 100.0] | 21.7 [-115.4 to 100.0]
  Transition Phase, n=68, 66, 20 | 73.1 [-90.5 to 100.0] | 100.0 [-100.0 to 100.0] | 100.0 [-100.0 to 100.0]
  Open-Label Phase, n=68, 64, 23 | 89.2 [-116.7 to 100.0] | 95.0 [-100.0 to 100.0] | 31.7 [-194.7 to 100.0]
  Last 8 weeks of Open-Label Phase, n=68, 63, 19 | 100.0 [-184.2 to 100.0] | 100.0 [-53.3 to 100.0] | 100.0 [-500.0 to 100.0]

9. Secondary Outcome: Number of Participants With >=25%, >=50%, >=75%, or 100% Reduction or >=50% Increase From Baseline in Weekly PGTC Seizure Frequency for the Entire Continuation Phase, the Transition Phase, the Open-Label (OL) Phase, and the Last 8 Weeks of the OL Phase.
Description: Change in seizure frequency was calculated as the average seizure frequency during each of the following: the Entire CP (CP Week 1 up to Week 52); the Transition Phase (CP Week 1 up to Week 7); the Open-Label (OL) Phase (CP Week 8 up to Week 52); and the last 8 weeks of the Open Label Phase (CP Week 45 up to Week 52) minus the seizure frequency at Baseline. W, Week.
Time Frame: as for outcome 8
Population: ITT Population for CP. Variability in participant numbers are due to not having any PGTC seizures during the Baseline Phase and study withdrawal prior to progressing to the next phase.
Measure: Number; unit: participants
Arm/Group | Continuation Phase: Placebo/LTG | Continuation Phase: LTG/LTG | Baseline Failures
Number analyzed (Participants) | 68 | 66 | 24
participants
  >=25% reduction, Entire CP, n=68, 66, 24 | 59 | 63 | 11
  >=50% reduction, Entire CP, n=68, 66, 24 | 57 | 59 | 11
  >=75% reduction, Entire CP, n=68, 66, 24 | 46 | 49 | 8
  100% reduction, Entire CP, n=68, 66, 24 | 16 | 28 | 6
  >=50% increase, Entire CP, n=68, 66, 24 | 2 | 1 | 10
  >=25% reduction, Transition Phase, n=68, 66, 20 | 51 | 60 | 13
  >=50% reduction, Transition Phase, n=68, 66, 20 | 44 | 56 | 12
  >=75% reduction, Transition Phase, n=68, 66, 20 | 33 | 46 | 12
  100% reduction, Transition Phase, n=68, 66, 20 | 27 | 41 | 12
  >=50% increase, Transition Phase, n=68, 66, 20 | 3 | 1 | 3
  >=25% reduction, Open-Label Phase, n=68, 64, 23 | 61 | 61 | 12
  >=50% reduction, Open-Label Phase, n=68, 64, 23 | 56 | 57 | 10
  >=75% reduction, Open-Label Phase, n=68, 64, 23 | 47 | 49 | 8
  100% reduction, Open-Label Phase, n=68, 64, 23 | 21 | 28 | 6
  >=50% increase, Open-Label Phase, n=68, 64, 23 | 2 | 1 | 10
  >=25% reduction, Last 8 W of OL Phase,n=68, 63, 19 | 60 | 60 | 10
  >=50% reduction, Last 8 W of OL Phase,n=68, 63, 19 | 53 | 53 | 10
  >=75% reduction, Last 8 W of OL Phase,n=68, 63, 19 | 45 | 47 | 10
  100% reduction, Last 8 W of OL Phase, n=68, 63, 19 | 35 | 41 | 10
  >=50% increase, Last 8 W of OL Phase, n=68, 63, 19 | 2 | 1 | 4

10. Secondary Outcome: Mean Change From Baseline in the Profile of Mood State (POMS) Mood Disturbance Total Score at Week 19 of the Double-Blind Treatment Phase
Description: The POMS is a self-administered 65-item questionnaire that evaluates the participants' perception of their mood state in 6 areas: tension-anxiety, depression-dejection, anger-hostility, vigor-activity, fatigue-inertia, and confusion-bewilderment. Items are rated on a 5-point Likert scale from 0 (not at all) to 4 (extremely), with higher scores indicating a more negative mood state. A total score (from 0 to 24) is obtained by summing the scores of the six domains.
Time Frame: Baseline and Week 19 (or last on-study measurement in Double-Blind Treatment Phase)
Population: ITT Population. The questionnaire was not completed by 53 and 57 participants in the Placebo and LTG XR groups, respectively. Only participants completing the questionnaire were included in the analysis of this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: LTG XR
Number analyzed (Participants) | 20 | 13
points on a scale | 2.4 (6.97) | 9.7 (8.65)

11. Secondary Outcome: Mean Change From Baseline in the Center for Epidemiological Studies-Depression Scale (CES-D) Total Score at Week 19 of the Double-Blind Treatment Phase
Description: The 20-item CES-D questionnaire is self-administered and asks respondents to report the frequency to which the 20 events were experienced over the past week. A 4-point Likert scale is used and ranges from rarely or none of the time (0) to most or all of the time (3). The total score, a sum across the 20 items (ranging from 0 to 60), determines the extent to which a participant may be experiencing depression. Higher scores indicate a higher severity of depression.
Time Frame: Baseline and Week 19 (or last on-study measurement in Double-Blind Treatment Phase)
Population: ITT Population. The questionnaire was not completed by 64 and 59 participants in the Placebo and LTG XR groups, respectively. Only participants completing the questionnaire were included in the analysis of this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: LTG XR
Number analyzed (Participants) | 9 | 11
points on a scale | 2.9 (2.81) | 2.4 (2.54)

12. Secondary Outcome: Mean Change From Baseline in the Neurological Disorders Depression Inventory-Epilepsy (NDDI-E) 6-Item Total Score at Week 19 of the Double-Blind Treatment Phase
Description: The NDDI-E is a self-reported questionnaire composed of 46 brief phrases/words to identify mood disorders across the spectrum of depression. It was developed to capture depressive moods that are co-morbid with the disease of epilepsy or its treatment as well as to measure the depressive state of the participant. All phrases are measured on a 4-point Likert scale of Never (1) to Always/often (4) and refer to the participants' mood over the past week. Scoring is comprised of a total mood score calculated by summing the scores of 6 specific items (from 6=never to 24=always or often).
Time Frame: Baseline and Week 19 (or last on-study measurement in Double-Blind Treatment Phase)
Population: ITT Population. The questionnaire was not completed by 65 participants in both the Placebo and LTG XR groups. Only participants completing the questionnaire were included in the analysis of this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: LTG XR
Number analyzed (Participants) | 8 | 5
points on a scale | -0.1 (0.98) | -2.4 (1.24)

13. Secondary Outcome: Mean Change From Baseline in the Quality of Life in Epilepsy-31-P (QOLIE-31P) Overall Score at Week 19 of the Double-Blind Treatment Phase
Description: The QOLIE-31 is a 31-item questionnaire that evaluates the participants' perception of his or her quality of life in 7 domains: seizure worry, emotional well being, energy/fatigue, cognitive functioning, medication effects, social functioning, and overall quality of life. Each domain (with scores ranging from 0 to 100) is summed and divided by the total number of questions that were answered. The overall score is derived by weighting and then summing up the seven domain scores.
Time Frame: Baseline and Week 19 (or last on-study measurement in Double-Blind Treatment Phase)
Population: ITT Population. The questionnaire was not completed by 55 participants in both the Placebo and LTG XR groups. Only participants completing the questionnaire were included in the analysis of this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: LTG XR
Number analyzed (Participants) | 18 | 15
points on a scale | -6.5 (3.97) | -8.5 (4.35)

14. Secondary Outcome: Mean Change From Baseline in the Adverse Experience Profile (AEP) Total Score at Week 19 of the Double-Blind Treatment Phase
Description: The AEP is a list of 19 items covering many possible side effects attributable to drug treatment. The participants respond by assessing how much each event has been a problem for them over the past 4 weeks (1=Never a Problem to 4=Always a Problem). Each individual item can be examined; an overall adverse events score is calculated as the sum of the scores across the 19 items. The AEP total score ranges from 19 to 76, with a higher score indicating a higher degree of adverse event severity.
Time Frame: Baseline and Week 19 (or last on-study measurement in Double-Blind Treatment Phase)
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: LTG XR
Number analyzed (Participants) | 8 | 5
points on a scale | 3.0 (2.16) | 1.4 (2.77)

15. Secondary Outcome: Mean Change From Baseline in the Seizure Severity Questionnaire (SSQ) Global Bother Score at Week 19 Double-Blind Treatment Phase
Description: The SSQ is a self-reported instrument developed to assess the severity of seizures and seizure symptoms. The scale consists of 10 major clinical features/symptoms of seizures that the participants rate on a 7-point Likert scale (ranging from very mild/helpful/no bother at all [1] to very severe/no help/bothersome [7]). The Global Bother Domain is the primary score used for the analysis of the SSQ and has scores ranging from 1 to 7.
Time Frame: Baseline and Week 19 (or last on-study measurement in Double-Blind Treatment Phase)
Population: ITT Population. The questionnaire was not completed by 68 and 67 participants in the Placebo and LTG XR groups, respectively. Only participants completing the questionnaire were included in the analysis of this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: LTG XR
Number analyzed (Participants) | 5 | 3
points on a scale | 0.86 (0.84) | 1.23 (1.08)

16. Secondary Outcome: Mean Change From Baseline in the Epworth Sleepiness Scale (ESS) 8-Item Total Score at Week 19 of the Double-Blind Treatment Phase
Description: The ESS is an 8-item, self-administered questionnaire that measures excessive daytime sleepiness in adults. The instrument captures information on the extent to which the participant would be likely, or not, to fall asleep in certain situations. The stimulus question is: How likely are you to doze off or fall asleep in the following situations, in contrast to feeling just tired? Questions are answered on a 4-point scale (would never doze [0] to high chance of dozing [3]). The total score ranges from 0 to 24, where a higher score indicates a higher chance of dozing.
Time Frame: Baseline and Week 19 (or last on-study measurement in Double-Blind Treatment Phase)
Population: ITT Population. The questionnaire was not completed by 55 and 51 participants in the Placebo and LTG XR groups, respectively. Only participants completing the questionnaire were included in the analysis of this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: LTG XR
Number analyzed (Participants) | 18 | 19
points on a scale | -0.6 (0.69) | 1.0 (0.67)

17. Secondary Outcome: Serum Concentrations and Population (POP) Pharmacokinetic Parameters for Lamotrigine
Description: Serum samples for participants on lamotrigine were analyzed with a validated analytical method based on solid phase extraction of serum followed by High-Performance Liquid Chromatography (HPLC) Mass Spectrometry (MS)/MS analysis. The lower limit of quantification (LLQ) for serum lamotrigine was 4 nanograms (ng)/milliliter (mL), using a 50 microliter (µL) aliquot of human serum with a higher limit of quantification (HLQ) of 4,000 ng/mL. PK data cannot be reported, as PK data from several different studies have been combined into one POP/PK analysis and cannot be separated by study.
Time Frame: Blood samples drawn at Treatment Weeks 11, 15, and 19 (or last on-study measurement in Double-Blind Treatment Phase)
Population: PK Population: Number of participants analyzed for PK data cannot be reported, as PK data from several different studies have been combined into one POP/PK analysis and cannot be separated by study.
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: LTG XR
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Serious adverse events (SAEs) and adverse events (AEs) were collected for all participants in the Safety Population. The Safety Population was defined as all participants who took at least one dose of study drug.
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: LTG XR | Continuation Phase: Placebo/LTG | Continuation Phase: LTG/LTG | Baseline Failures
Serious Adverse Events (participants affected / at risk) | 0/74 | 1/72 | 3/69 | 3/67 | 1/32
Other Adverse Events (participants affected / at risk) | 21/74 | 27/72 | 29/69 | 21/67 | 18/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Phase: Placebo (N=74) | Double-Blind Phase: LTG XR (N=72) | Continuation Phase: Placebo/LTG (N=69) | Continuation Phase: LTG/LTG (N=67) | Baseline Failures (N=32)
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope vasovagal (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Conversion disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Phase: Placebo (N=74) | Double-Blind Phase: LTG XR (N=72) | Continuation Phase: Placebo/LTG (N=69) | Continuation Phase: LTG/LTG (N=67) | Baseline Failures (N=32)
Headache (Nervous system disorders) | 12 | 10 | 11 | 5 | 9
Dizziness (Nervous system disorders) | 5 | 4 | 7 | 4 | 7
Tremor (Nervous system disorders) | 0 | 4 | 5 | 3 | 3
Vomiting (Gastrointestinal disorders) | 3 | 7 | 5 | 2 | 2
Nausea (Gastrointestinal disorders) | 4 | 5 | 1 | 1 | 5
Pyrexia (General disorders) | 4 | 5 | 7 | 5 | 3
All rash (Skin and subcutaneous tissue disorders) | 4 | 2 | 2 | 1 | 2
Diplopia (Eye disorders) | 1 | 4 | 4 | 1 | 2
Ataxia (Nervous system disorders) | 0 | 0 | 2 | 2 | 2
Somnolence (Nervous system disorders) | 0 | 1 | 1 | 2 | 2
Pain (General disorders) | 2 | 2 | 3 | 2 | 2
Fatigue (General disorders) | 2 | 1 | 1 | 0 | 3
Nasopharyngitis (Infections and infestations) | 1 | 2 | 4 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 2
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.